CLINICAL TRIAL: NCT02795091
Title: Comparision of Different Methods of Enviromennt Disinfection
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chun Pan (Other)
Responsible Party: Sponsor-Investigator, Chun Pan, doctor, Southeast University, China
Organization: Southeast University, China (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: enviromennt disinfection
Record Dates: First submitted 2016-06-05; First posted 2016-06-09 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Enviroment Cleaning
Keywords: clean supplies; ICU floor; bacteria colony; catheter associated with infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual clean (Other): clean the rag and floor towel manually
  Interventions: Other: manual cleaning
- machine clean (Other): clean the rag and floor towel by machine
  Interventions: Device: machine clean

INTERVENTIONS:
Other: manual cleaning — manual clean the rag and floor towel
  Arms: Manual clean
Device: machine clean — machine clean the rag and floor towel
  Arms: machine clean

SUMMARY:
Multidrug resistance bacteria infection is common in ICU. Infection incidence is associated with age, organ dysfunction, invasive treatment and enviroment cleaning. According to hospital hygienic standard for disinfection, total numbers of colony of air and the object surface in ICU must be ≤4CFU/cm2（5min）and≤10CFU/cm2. in this study, the two different methods will be used to evaluate the disinfection effects in ICU enviroments.

ELIGIBILITY:
Inclusion Criteria:

no patients recruitment

Exclusion Criteria:

no patients recruitment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
incidence of infection | up to one month

SECONDARY OUTCOMES:
dose of antibiotics | up to one month

IPD SHARING:
Plan to Share IPD: Undecided